CLINICAL TRIAL: NCT00340171
Title: Fetal Growth Evaluation by Three-Dimensional Ultrasound
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999997068; OH97-CH-N068
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Pregnancy
Keywords: Intrauterine Growth Retardation; Natural History
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

GROUPS / COHORTS (1):
- Pregnant women and infants: pregnant women with singleton pregnancy and their newborns

SUMMARY:
Fetal growth abnormalities, such as macrosomia and intrauterine growth retardation, are an important cause for increased perinatal mortality in the United States. Toward this end, accurate fetal weight determinations are very important for guiding prenatal care. Three-dimensional ultrasound is a recent technology that provides a new way to evaluate the fetus. This technique allows one to arbitrarily scan through a digital ultrasound volume dataset, visualize organs from different perspectives, and render anatomical features through computer processing. It also allows the retrospective measurement of distances and volumes even in the physical absence of the patient.

A maximum of 400 pregnancies will be serially studied by three-dimensional ultrasound to characterize the growth of volume parameters such as the fetal thigh. This information will be applied to the Rossavik model of individualized growth assessment. The technique allows growth evaluation by comparing various ultrasound measurements or birth characteristics to the individual growth standards specified by the prediction model. Newborn infant body composition will also be studied within 48 hours of delivery.

A separate cross-sectional study of up to 2,577 fetuses will allow development of birth weight prediction models based upon fetal volume measurements and further analysis of fetal growth abnormalities. Individual growth curve standards utilizing these volume parameters should allow one to evaluate deviations from expected growth or birth weight by using each fetus as its own control.

DETAILED DESCRIPTION:
Fetal growth abnormalities, such as macrosomia and intrauterine growth retardation, are an important cause for increased perinatal mortality in the United States. Toward this end, accurate fetal weight determinations are very important for guiding prenatal care. Three-dimensional ultrasound is a recent technology that provides a new way to evaluate the fetus. This technique allows one to arbitrarily scan through a digital ultrasound volume dataset, visualize organs from different perspectives, and render anatomical features through computer processing. It also allows the retrospective measurement of distances and volumes even in the physical absence of the patient.

This protocol consists of two study arms and emphasizes the ability of 3D ultrasound to reliably measure fetal soft tissue as an index of generalized nutritional status. The longitudinal arm will enroll 400 pregnancies to allow the use of 2D and 3D ultrasonography for characterizing serial growth patterns of sonographic parameters throughout pregnancy. This approach compares ultrasound measurements or birth characteristics to individual growth standards specified by Rossavik prediction models. After delivery, a maximum of 329 newborn infants, resulting from the same pregnancies, will have correlative photographs and measurements of their head, abdomen, thigh, skin folds, weight, and crown-heel length taken to classify growth outcome. Noninvasive air displacement plethymography will be used to measure neonatal percent body fat and lean body mass after delivery. Infant body composition data will allow the precise classification of neonatal growth outcome for subsequent correlation to prenatal sonographic studies. The cross-sectional arm of this protocol will allow sonographic studies of 2,577 fetuses with similar correlative neonatal evaluation of 1,212 infants for a total of 3,789 subjects. The results will be used to develop a new fetal weight estimation models that combine 2D and 3D sonographic parameters to improve accuracy and precision of these predictions. A maximum of 50 newborns from this cross-sectional arm will also be re-evaluated for infant body composition at 1 and 2 weeks following delivery to document changes in percent body fat and fat-free mass. Therefore, the subject recruitment ceiling would be (2,577 mothers + 1,212 infants) + (400 mothers + 329 infants) or 4,518 total subjects for this Protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

ALL SUBJECTS:

Pregnant women between the ages of 18 and 40 years at Hutzel and William Beaumont Hospital sites.

LOGITUDINAL ARM:

Single gestation.

No pregnancy complications.

Accurate dating criteria (sure LMP or first trimester scan).

CROSS-SECTIONAL ARM OF PROTOCOL:

Singe Gestation.

No pregnancy complications.

Accurate data criteria (sure LMP or 1st trimester scan).

Delivery anticipated within 4 days of scan.

INFANT BODY COMPOSITION STUDY

Birthweight above 1,000 grams

EXCLUSION CRITERIA:

LONGITUDINAL ARM OF PROTOCOL:

Poor visualization of the fetus due to technical factors (e.g. obesity).

Risk factors that increase risk for not keeping serial ultrasound appointments.

CROSS-SECTIONAL ARM OF PROTOCOL:

Poor visualization of the fetus due to technical factors (e.g. obesity).

Hemodynamically unstable patients.

INFANT BODY COMPOSITION STUDY

Infants requiring mechanical ventilation, heart monitors, or intravenous fluid.

Hemodynamically unstable infant

Infants with thermoregulation problems

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women aged 18 years and older attending clinics at the Hutzel Women's Hospital in Detroit.
Sampling Method: Non-Probability Sample
Enrollment: 1919 (Actual)
Dates: Start 1997-12-04 (Actual); Primary Completion 2012-11-05 (Actual); Study Completion 2012-11-05 (Actual)

PRIMARY OUTCOMES:
Intrauterine fetal growth restriction | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Romero, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (2):
- United States (2):
  - Hutzel Women's Hospital, Detroit, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan